CLINICAL TRIAL: NCT03034460
Title: Efficacy and Safety of CD5024 1% in Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RD.03.SPR.109807
Record Dates: First submitted 2016-11-21; First posted 2017-01-27 (Estimated); Results first posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2017-01

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- CD5024 1% cream (Experimental): Active drug;
  Interventions: Drug: CD5024 1% cream
- CD5024 cream placebo (Placebo Comparator): Placebo of active drug;
  Interventions: Drug: CD5024 cream placebo
- CD0271/CD1579 gel (Other): Positive control;
  Interventions: Drug: CD0271/CD1579 gel
- CD0271/CD1579 gel placebo (Other): Placebo of positive control;
  Interventions: Drug: CD0271/CD1579 gel placebo

INTERVENTIONS:
Drug: CD5024 1% cream — 500 µL on half-face, five days a week during 6 weeks
  Arms: CD5024 1% cream
Drug: CD5024 cream placebo — 500 µL on half-face, five days a week during 6 weeks
  Arms: CD5024 cream placebo
Drug: CD0271/CD1579 gel — 500 µL on half-face, five days a week during 6 weeks
  Arms: CD0271/CD1579 gel
Drug: CD0271/CD1579 gel placebo — 500 µL on half-face, five days a week during 6 weeks
  Arms: CD0271/CD1579 gel placebo

SUMMARY:
Exploratory, multi-center, randomised, investigator-blinded, vehicle controlled study using intra-individual comparison involving subjects with acne vulgaris on face to evaluate the efficacy of CD5024 1% cream over a 6-week treatment period compared to its vehicle.

DETAILED DESCRIPTION:
Study drugs application will be performed once daily, 5 days a week during 6 weeks

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a male or a female aged from 18 to 35 years old at screening visit.
2. The subject has a medical diagnosis of acne vulgaris :

   2.1 at least 20 (twenty) inflammatory lesions and a maximum of 100 (one hundred) non-inflammatory lesions (nose is excluded for the lesion count) at Baseline

   2.2 symmetry of the lesions: No more than twice as many acne lesions on one side as compared to the other side at Baseline
3. If the subject is a female of childbearing potential, she must agree to use an effective contraceptive method for the duration of the study

Exclusion Criteria:

1. The subject has an underlying known disease surgical or medical condition, in the opinion of the investigator might interfere with interpretation of the study results or put the subject at risk (e.g., other dermatological diseases affecting the treatment area, such as a dermatitis, eczema, etc., or any uncontrolled chronic or serious diseases which would normally prevent participation in any clinical study, such as a cancer, leukemia or severe hepatic impairment), (Screening).
2. The subject has acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne, etc.), nodulo cystic acne, or acne requiring systemic treatment.
3. The subject has a known or suspected allergies or sensitivities to any components of any of the study drugs (see Investigator's Brochure/Product label).
4. The subject is a male with beard or facial hair, which would interfere with clinical evaluation or clinical procedure (Screening and Baseline).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2016-11-02 (Actual); Study Completion 2016-11-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (2):
  - Galderma Investigational Site (# 8060), Windsor, Ontario
  - Galderma Investigational site, Montreal, Quebec
- France (2):
  - Galderma investigational site, Nantes
  - Galderma investigational site, Nice
- Germany (3):
  - Galderma investigational site, Berlin
  - Galderma investigational site, Bochum
  - Galderma investigational site, Münster

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at six centers in three countries (Germany, France, Canada) between 25 April 2016 (first participant screened) to 02 November 2016 (last participant completed).
Pre-assignment Details: A total of 70 participants were randomized, of which 64 participants completed the study.
Groups:
- Group I: CD5024 Cream Versus Its Vehicle: Participants applied 500 microliter (mcL) of CD5024 1% cream on one side of the face and matching placebo cream on the other side of the face once daily for 5 days a week from Week 1 to Week 5 and 4 days during Week 6 for a total of 29 applications.
- Group II: Epiduo Gel Versus Its Vehicle: Participants applied 500 mcL of Adapalene benzoyl peroxyde (Epiduo) gel on one side of the face and matching placebo cream on the other side of the face once daily for 5 days a week from Week 1 to Week 5 and 4 days during Week 6 for a total of 29 applications.
Period: Overall Study
Arm/Group | Group I: CD5024 Cream Versus Its Vehicle | Group II: Epiduo Gel Versus Its Vehicle
Started | 48 | 22
Completed | 45 | 19
Not Completed | 3 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Personal Reasons | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I: CD5024 Cream Versus Its Vehicle | Group II: Epiduo Gel Versus Its Vehicle | Total
Number analyzed (Participants) | 48 | 22 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.3 (4.7) | 23.4 (4.4) | 23.3 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 14 | 48
  Male | 14 | 8 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 46 | 14 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Number of inflammatory lesions [Mean (Standard Deviation); unit: Lesion Count] | 34.0 (11.6) | 34.2 (15.1) | 34.0 (12.7)

OUTCOME MEASURES:

1. Primary Outcome: Inflammatory Lesion Count (Papules and Pustules) at Day 40
Description: Inflammatory lesion count corresponded to the sum of papules and pustules.
Time Frame: Day 40
Population: This analysis was performed on ITT- last observation carried forward (LOCF) population. ITT-population included all participants who were randomized. Outcome measure data was summarized using the LOCF at Day 40. The data was planned, analyzed and reported for active (cream/gel) application on one side of face and vehicle controlled (matched cream/gel) on other side of face.
Measure: Mean (Standard Deviation); unit: lesion count
Units Other Than Participants: One side of face
Groups:
- CD5024 1% Cream: Participants applied CD5024 1% cream once daily for 5 days a week from Week 1 to Week 5 and for 4 days during Week 6.
- CD5024 1% Cream Matched Placebo: Participants applied CD5024 1% cream matched placebo once daily for 5 days a week from Week 1 to Week 5 and for 4 days during Week 6.
- Adapalene Benzoyl Peroxyde: Participants applied Adapalene Benzoyl Peroxyde once daily for 5 days a week from Week 1 to Week 5 and for 4 days during Week 6.
- Adapalene Benzoyl Peroxyde Matched Placebo: Participants applied Adapalene Benzoyl Peroxyde matched placebo once daily for 5 days a week from Week
  1 to Week 5 and for 4 days during Week 6.
Arm/Group | CD5024 1% Cream | CD5024 1% Cream Matched Placebo | Adapalene Benzoyl Peroxyde | Adapalene Benzoyl Peroxyde Matched Placebo
Number analyzed (Participants) | 48 | 48 | 22 | 22
Number analyzed (One side of face) | 48 | 48 | 22 | 22
lesion count | 10.1 (5.8) | 8.9 (5.0) | 6.1 (4.9) | 9.4 (5.7)
Statistical Analysis 1: Comparison: CD5024 1% Cream vs CD5024 1% Cream Matched Placebo; This analysis was performed in participants applied CD5024 1% Cream on one side of face and CD5024 1% Cream Matched Placebo on other side of face for paired difference between Active - Vehicle (CD5024 1% Cream [n=48] versus CD5024 1% Cream Matched Placebo [n=48]); Test type: Superiority; p = 0.158, Wilcoxon rank signed test
Statistical Analysis 2: Comparison: Adapalene Benzoyl Peroxyde vs Adapalene Benzoyl Peroxyde Matched Placebo; This analysis was performed in participants applied Adapalene Benzoyl Peroxyde on one side of face and Adapalene Benzoyl Peroxyde Matched Placebo on the other side of face for paired difference between Active - Vehicle (Adapalene Benzoyl Peroxyde [n=22] versus Adapalene Benzoyl Peroxyde Matched Placebo [n=22]); Test type: Superiority; p = 0.002, Wilcoxon rank signed test

2. Secondary Outcome: Inflammatory Lesion Count (Papules and Pustules) at Baseline (Day 1)
Description: Inflammatory lesion count corresponded to the sum of papules and pustules.
Time Frame: Baseline (Day 1)
Population: This analysis was performed on ITT population. ITT population included all partcipants who were randomized. The data was planned, analyzed and reported for active (cream/gel) application on one side of face and vehicle controlled (matched cream/gel) on other side of face.
Measure: Mean (Standard Deviation); unit: lesion count
Units Other Than Participants: One side of face
Arm/Group | CD5024 1% Cream | CD5024 1% Cream Matched Placebo | Adapalene Benzoyl Peroxyde | Adapalene Benzoyl Peroxyde Matched Placebo
Number analyzed (Participants) | 48 | 48 | 22 | 22
Number analyzed (One side of face) | 48 | 48 | 22 | 22
lesion count | 16.5 (4.9) | 17.5 (7.4) | 17.6 (8.6) | 16.6 (7.2)

3. Secondary Outcome: Percent Reduction From Baseline (Day 1) in Inflammatory Lesion Count at Day 40
Description: Inflammatory lesion count corresponded to the sum of papules and pustules.
Time Frame: Baseline (Day 1), and Day 40
Population: This analysis was performed on ITT population. ITT population included all participants who were randomized. The data was planned, analyzed and reported for active (cream/gel) application on one side of face and vehicle controlled (matched cream/gel) on other side of face.
Measure: Mean (Standard Deviation); unit: percent reduction of lesion count
Units Other Than Participants: One side of face
Arm/Group | CD5024 1% Cream | CD5024 1% Cream Matched Placebo | Adapalene Benzoyl Peroxyde | Adapalene Benzoyl Peroxyde Matched Placebo
Number analyzed (Participants) | 48 | 48 | 22 | 22
Number analyzed (One side of face) | 48 | 48 | 22 | 22
percent reduction of lesion count | 35.7 (43.4) | 44.4 (32.3) | 65.5 (24.0) | 42.5 (30.1)

4. Secondary Outcome: Total Lesion Count at Baseline (Day 1) and Day 40
Description: Total lesion counts corresponded to the sum of inflammatory and non-inflammatory lesions, and papules.
Time Frame: Baseline (Day 1), and Day 40
Population: This analysis was performed on ITT- last observation carried forward (LOCF) population. ITT population included all participants who were randomized. Outcome Measure data was summarized using the LOCF at Day 40. The data was planned, analyzed and reported for active (cream/gel) application on one side of face and vehicle controlled (matched cream/gel) on other side of face.
Measure: Mean (Standard Deviation); unit: lesion count
Units Other Than Participants: One side of face
Arm/Group | CD5024 1% Cream | CD5024 1% Cream Matched Placebo | Adapalene Benzoyl Peroxyde | Adapalene Benzoyl Peroxyde Matched Placebo
Number analyzed (Participants) | 48 | 48 | 22 | 22
Number analyzed (One side of face) | 48 | 48 | 22 | 22
lesion count
  Baseline (Day 1) | 37.7 (11.2) | 39.4 (13.7) | 37.3 (20.2) | 36.4 (18.0)
  Day 40 | 26.4 (16.8) | 25.9 (14.3) | 19.3 (15.0) | 25.5 (17.2)

5. Secondary Outcome: Percent Reduction From Baseline (Day 1) in Total Lesions at Day 40
Description: Total lesion counts corresponded to the sum of inflammatory and non-inflammatory lesions, and papules.
Time Frame: Baseline (Day 1), and Day 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent reduction in total lesion count
Units Other Than Participants: One side of face
Arm/Group | CD5024 1% Cream | CD5024 1% Cream Matched Placebo | Adapalene Benzoyl Peroxyde | Adapalene Benzoyl Peroxyde Matched Placebo
Number analyzed (Participants) | 48 | 48 | 22 | 22
Number analyzed (One side of face) | 48 | 48 | 22 | 22
percent reduction in total lesion count | 32.5 (32.2) | 34.0 (27.1) | 50.2 (27.2) | 27.8 (31.8)

6. Secondary Outcome: Non-Inflammatory Lesion Count at Baseline (Day 1) and Day 40
Description: Non-inflammatory lesion counts corresponded to the sum of open and closed comedones.
Time Frame: Baseline (Day 1), and Day 40
Population: as for outcome 3
Measure: Mean (Standard Error); unit: lesion count
Units Other Than Participants: One side of face
Arm/Group | CD5024 1% Cream | CD5024 1% Cream Matched Placebo | Adapalene Benzoyl Peroxyde | Adapalene Benzoyl Peroxyde Matched Placebo
Number analyzed (Participants) | 48 | 48 | 22 | 22
Number analyzed (One side of face) | 48 | 48 | 22 | 22
lesion count
  Baseline (Day 1) | 21.1 (9.5) | 21.8 (10.7) | 19.6 (14.1) | 19.6 (13.6)
  Day 40 | 16.2 (13.1) | 16.9 (12.7) | 13.0 (12.0) | 16.0 (14.1)

7. Secondary Outcome: Percent Reduction From Baseline in Non-Inflammatory Lesion at Day 40
Description: Non-inflammatory lesion counts corresponded to the sum of open and closed comedones.
Time Frame: Baseline (Day 1), and Day 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent reduction of lesion count
Units Other Than Participants: One side of face
Arm/Group | CD5024 1% Cream | CD5024 1% Cream Matched Placebo | Adapalene Benzoyl Peroxyde | Adapalene Benzoyl Peroxyde Matched Placebo
Number analyzed (Participants) | 48 | 48 | 22 | 22
Number analyzed (One side of face) | 48 | 48 | 22 | 22
percent reduction of lesion count | 27.8 (39.4) | 21.3 (42.0) | 36.9 (36.1) | 11.7 (48.6)

8. Secondary Outcome: Number of Participants Reported for Investigator's Preference on a 5-Point Scale at Day 40
Description: The Investigator gave opinion on their preference after comparison of the left and right sides of the face using the 5-point scale ranging from -2 to 2. The score and description indicated as follows: -2= left side of the face much better than right side, -1= left side of the face better than right side, 0= no clinical difference between the right and left sides of the face, 1= right side of the face better than the left side, 2= right side of the face much better than the left side.
Time Frame: Day 40
Population: This analysis was performed on ITT population. ITT population included all participants who were randomized. Here 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I: CD5024 Cream Versus Its Vehicle | Group II: Epiduo Gel Versus Its Vehicle
Number analyzed (Participants) | 48 | 48
Participants
  Day 40 (Active much better than Vehicle) | 0 | 4
  Day 40 (Active better than Vehicle) | 16 | 7
  Day 40 (No clinical difference between Active and Vehicle) | 16 | 6
  Day 40 (Vehicle better than Active) | 14 | 4
  Day 40 (Vehicle much better than Active) | 1 | 0

9. Secondary Outcome: Number of Participants Reported for Participant's Preference on 5-Point Scale at Day 40
Description: The participants gave opinion on their preference after comparison of the left and right sides of the face using the 5-point scale ranging from -2 to 2. The score and description indicated as follows: -2= left side of the face much better than right side, -1= left side of the face better than right side, 0= no clinical difference between the right and left sides of the face, 1= right side of the face better than the left side, 2= right side of the face much better than the left side.
Time Frame: Day 40
Population: This analysis was performed on ITT population. ITT population included all participants who were randomized. Here 'N' (number of participants analyzed) signifies participants who were evaluable for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I: CD5024 Cream Versus Its Vehicle | Group II: Epiduo Gel Versus Its Vehicle
Number analyzed (Participants) | 47 | 21
Participants
  Day 40 (Active much better than Vehicle) | 2 | 2
  Day 40 (Active better than Vehicle) | 11 | 11
  Day 40 (No clinical difference between Active and Vehicle) | 15 | 4
  Day 40 (Vehicle better than Active) | 16 | 3
  Day 40 (Vehicle much better than Active) | 3 | 1

10. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: AE was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily had a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory value), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From start of study up to follow up (Week 7)
Population: This analysis was performed on safety population. Safety population included participants in the ITT population who received at least 1 application of the investigational product. Number of participants with AE's were reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I: CD5024 Cream Versus Its Vehicle | Group II: Epiduo Gel Versus Its Vehicle
Number analyzed (Participants) | 48 | 22
Participants | 32 | 14

11. Secondary Outcome: Number of Participants Reported Worst Local Tolerability Score on Treated Areas (Face and Ear) From Day 1 to Follow up (Week 7)
Description: Signs and symptoms of local cutaneous irritation(local tolerability [erythema, scaling, dryness, stinging/burning, pruritus]) were evaluated on all treated areas (face and behind ears if applicable) every day from Day 1 up to follow-up (Week 7) using a 4-point scale of None (0), Mild (1), Moderate (2), or Severe (3). Number of participants reported worst local tolerability score on treated areas from Day 1 to follow up (Week 7) was reported.
Time Frame: From Day 1 up Follow up (Week 7)
Population: Safety population included participants in the ITT population who received at least 1 application of the investigational product. Here 'n' (number analyzed) signifies number of participants who were evaluable for each specified category. The data was planned, analyzed and reported for active (cream/gel) application on one side of face and vehicle controlled (matched cream/gel) on other side of face.
Measure: Count of Participants; unit: Participants
Arm/Group | CD5024 1% Cream | CD5024 1% Cream Matched Placebo | Adapalene Benzoyl Peroxyde | Adapalene Benzoyl Peroxyde Matched Placebo
Number analyzed (Participants) | 48 | 48 | 22 | 22
Participants
  Face: Erythema: 0-None | 37 | 38 | 8 | 15
  Face: Erythema: 1-Mild | 9 | 9 | 11 | 6
  Face: Erythema: 2-Moderate | 2 | 1 | 3 | 1
  Face: Scaling/Desquamation: 0-None | 38 | 38 | 5 | 16
  Face: Scaling/Desquamation: 1-Mild | 10 | 10 | 13 | 5
  Face: Scaling/Desquamation: 2- Moderate | 0 | 0 | 4 | 1
  Face: Dryness: 0-None | 38 | 37 | 4 | 10
  Face: Dryness: 1-Mild | 10 | 11 | 13 | 12
  Face: Dryness: 2-Moderate | 0 | 0 | 5 | 0
  Face: Stinging/Burning: 0-None | 44 | 43 | 8 | 17
  Face: Stinging/Burning: 1-Mild | 3 | 4 | 8 | 5
  Face: Stinging/Burning: 2-Moderate | 1 | 1 | 6 | 0
  Ear: Erythema: 0-None: number analyzed (Participants) | 22 | 22 | 11 | 11
  Ear: Erythema: 0-None | 20 | 20 | 8 | 11
  Ear: Erythema: 1-Mild: number analyzed (Participants) | 22 | 22 | 11 | 11
  Ear: Erythema: 1-Mild | 2 | 2 | 2 | 0
  Ear: Erythema: 2-Moderate: number analyzed (Participants) | 22 | 22 | 11 | 11
  Ear: Erythema: 2-Moderate | 0 | 0 | 1 | 0
  Ear: Scaling/Desquamation: 0-None: number analyzed (Participants) | 22 | 22 | 11 | 11
  Ear: Scaling/Desquamation: 0-None | 22 | 22 | 7 | 11
  Ear: Scaling/Desquamation: 1-Mild: number analyzed (Participants) | 22 | 22 | 11 | 11
  Ear: Scaling/Desquamation: 1-Mild | 0 | 0 | 3 | 0
  Ear: Scaling/Desquamation: 2-Moderate: number analyzed (Participants) | 22 | 22 | 11 | 11
  Ear: Scaling/Desquamation: 2-Moderate | 0 | 0 | 1 | 0
  Ear: Dryness: 0-None: number analyzed (Participants) | 22 | 22 | 11 | 11
  Ear: Dryness: 0-None | 22 | 22 | 7 | 10
  Ear: Dryness: 1-Mild: number analyzed (Participants) | 22 | 22 | 11 | 11
  Ear: Dryness: 1-Mild | 0 | 0 | 3 | 1
  Ear: Dryness: 2-Moderate: number analyzed (Participants) | 22 | 22 | 11 | 11
  Ear: Dryness: 2-Moderate | 0 | 0 | 1 | 0
  Ear: Stinging/Burning: 0-None: number analyzed (Participants) | 22 | 22 | 11 | 11
  Ear: Stinging/Burning: 0-None | 22 | 22 | 8 | 11
  Ear: Stinging/Burning: 1-Mild: number analyzed (Participants) | 22 | 22 | 11 | 11
  Ear: Stinging/Burning: 1-Mild | 0 | 0 | 2 | 0
  Ear: Stinging/Burning: 2-Moderate: number analyzed (Participants) | 22 | 22 | 11 | 11
  Ear: Stinging/Burning: 2-Moderate | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: From start of study up to follow up (Week 7)
Arm/Group | Group I: CD5024 Cream Versus Its Vehicle | Group II: Epiduo Gel Versus Its Vehicle
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/22
Other Adverse Events (participants affected / at risk) | 32/48 | 11/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I: CD5024 Cream Versus Its Vehicle (N=48) | Group II: Epiduo Gel Versus Its Vehicle (N=22)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 13 (13) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 14 (14) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes